CLINICAL TRIAL: NCT05641974
Title: Effect of Helpers Program On-line Training on Smoking Relapse and Social Networks
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-4624; 1R01CA248658-01A1 (NIH)
Record Dates: First submitted 2022-11-21; First posted 2022-12-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Smoking; Cigarette Smoking
Keywords: Smoking cessation; Relapse prevention
MeSH Terms: conditions — Smoking; Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician analyzing outcomes is blinded to study arm assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Helpers Stay Quit Training (Experimental): Research participants randomized to the experimental arm will receive the on-line Helpers Stay Quit training which provides training on how to help others quit smoking.
  Interventions: Behavioral: Helpers Stay Quit Training
- Usual Care (No Intervention): Research participants randomized to the arm without intervention will receive Quitline usual care. They will be contacted for assessment of abstinence at 7 months after enrollment in services. If the participant has relapsed, the Quitline will attempt to re-engage the participant in cessation services (telephone and/or web-based).

INTERVENTIONS:
Behavioral: Helpers Stay Quit Training — The Helpers Stay Quit training emphasizes a tobacco-user centered, non-confrontational approach to encouraging others to quit smoking. Helpers Stay Quit trainees learn how to offer a 4-step "helping conversation". The four steps of a helping conversation parallel the 4 core training modules of Helpers Stay Quit (Awareness, Understanding, Helping, Relating). A key learning objective of Helpers Stay Quit, is for Helpers to learn how to manage their own expectations for the process and outcome of a helping conversation (e.g. Helpers are taught that they cannot "make" anyone quit, but they can offer non-judgmental support, and information about effective cessation aids). Consequently, Helpers are taught to manage their own behavior when helping others (e.g. avoiding nagging or pushing a tobacco-user to quit). The helping conversation focuses on encouraging behavior change that is aligned with the tobacco user's current willingness/readiness to take any action toward quitting.
  Arms: Helpers Stay Quit Training

SUMMARY:
The purpose of this study is to assess the effect of the Helpers Stay Quit training on abstinence over time of newly abstinent smokers, and on the interactions they have with their personal network related to smoking and smoking cessation.

DETAILED DESCRIPTION:
Despite major gains in smoking cessation treatment, over half of recently quit smokers will relapse within the first year. To date, relapse prevention interventions have focused on the newly abstinent smoker ("abstainer"), and not attempted to directly or indirectly influence the abstainer's personal network, e.g. by helping the abstainer influence others in their personal network to quit. Personal networks exert powerful effects on initiating and maintaining smoking behavior, and can facilitate maintaining abstinence or trigger relapse. A "help others" intervention that seeks to increase the abstainer's ability to influence smokers in their personal network to quit - thereby creating a social environment more supportive of long-term abstinence - may have a beneficial effect on relapse. The Helpers Stay Quit intervention encourages abstainers to reinforce their own abstinence through helping others quit, and to proactively influence their personal network to be more conducive to long-term smoking abstinence. Helpers Stay Quit teaches abstainers how to encourage other tobacco users to quit and avoid relapse through a non-confrontational "helping conversation" that encourages quitting and use of evidence-based cessation aids (e.g. Quitlines, cessation medications) without confrontation and nagging. The investigator hypothesizes that Quitline abstainers exposed to Helpers Stay Quit will have higher 30-day and 7-day point prevalence abstinence than those receiving Quitline follow-up usual care, and that the effect of Helpers Stay Quit may be mediated by personal network characteristics. To test this hypothesis, the investigator proposes a pragmatic randomized controlled trial with embedded mixed-methods personal network study to assess the effect of Helpers Stay Quit training on proportion and duration of abstainers' abstinence over time, and on abstainer's personal network interactions related to smoking and smoking cessation. Metrics derived from the personal network study will be used for mediational analyses of overall, and gender-based effects of Helpers Stay Quit on smoking relapse.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Abstinent from smoking for between 14 and 60 days
* Primary tobacco use is cigarettes
* Has access to Internet via computer or mobile device
* Self-described proficiency with English
* Willing and able to send/receive weekly text messages using personal mobile phone plan
* Will allow Quitline to share their client data with research team
* Willing to complete online surveys at baseline, 3-, 6-, 9- and 12 months
* Willing to self-collect dried blood spot and send back to research team
* If assigned to Helpers Stay Quit condition, willing to complete training within 14 days
* If selected, willing to participate in qualitative interview
* Willing to forego any other training for tobacco cessation intervention/support (i.e., to become a cessation counselor/facilitator or support person, e.g., 'quit buddy') for the duration of their study enrollment

Exclusion Criteria:

* Any prior exposure to Helpers training or other cessation training in the previous 2 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 940 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
7-day and 30-day abstinence from using combustible tobacco at 6 months post-randomization | Self-reported data collected at 6 months post-randomization
  Participants report the number of days (if any) they smoked combustible tobacco within the specified timeframe.
7-day and 30-day abstinence from using combustible tobacco at 12 months post-randomization | Self-reported data collected at 12 months post-randomization
  Participants report the number of days (if any) they smoked combustible tobacco within the specified timeframe.

SECONDARY OUTCOMES:
7-day and 30-day abstinence from using combustible tobacco at 3 months and 9 months post-randomization | Self-reported data collected at 3- and 9-months post-randomization
  Participants report the number of days (if any) they smoked combustible tobacco within the specified timeframe.
Time to first relapse | Weekly data collected months 1-6, bi-weekly data collected months 7-12 post-randomization
  Participants report the number of days (if any) they smoked combustible tobacco within the specified timeframe.
Number, timing, and duration of relapses | Weekly data collected months 1-6, bi-weekly data collected months 7-12 post-randomization
  Participants report the number of days (if any) they smoked combustible tobacco within the specified timeframe.
Number of helping conversations offered | Weekly data collected months 1-6; bi-weekly data collected months 7-12; data collected at 3-, 6-, 9-, and 12-months post-randomization
  Participants report the number of helping conversations (if any) offered within the specified timeframe.
Biochemical confirmation of abstinence at 6 and 12 months on a subsample | Data collected and 6- and 12-months post-randomization
  Participants who report abstinence at 6- and 12-months (and no other exposure to nicotine) receive a dried blood spot kit which is returned and tested for cotinine.

CONTACTS AND LOCATIONS:
Overall Officials: Myra Muramoto, MD, MPH, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Muramoto ML, Hopkins A, Bell M, Allen A, Nair U, Connolly TE. Results of a Feasibility Study of Helpers Stay Quit Training for Smoking Relapse Prevention. Nicotine Tob Res. 2021 Mar 19;23(4):711-715. doi: 10.1093/ntr/ntaa176. PMID 32966558